CLINICAL TRIAL: NCT06217731
Title: Inflammatory Markers in Saliva of Patients With Burning Mouth Syndrome Before and After Treatment With Low-Level Laser Therapy and Clonazepam: A Randomized, Single-Blind Clinical Trial
Brief Title: Inflammatory Markers in Saliva of Patients With Burning Mouth Syndrome
Acronym: burningmouth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, Principal investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pia Lopez Jornet
Record Dates: First submitted 2024-01-06; First posted 2024-01-22 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-01

CONDITIONS: Burning Mouth Syndrome
Keywords: saliva; pain; markers
MeSH Terms: conditions — Burning Mouth Syndrome; Pain | interventions — Lasers; Clonazepam

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients who were included in Group 1 (n=20) were treated with the low power diode laser Helbo® Theralite Laser 3D Pocket Probe once a week for one month and Rivotril 0.25mg once every 24 hours for one month. Group 2 (n=19) were treated with the same laser once a week for one month, but with the tip not activated as a placebo treatment. Group 3 (n=21) were only treated with Helbo® laser once a week for one month and Group 4 (n=18) had only Rivotril 0.25mg once a day for one month. The patients were not aware of the different groups on which this study is based.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 laser + clonazepam (Active Comparator): Group 1 (n=20) were treated with the Helbo® Theralite Laser 3D Pocket Probe low power diode laser once a week for a month and Rivotril ( clonazepam) 0.25mg once every 24 hours for a month.
  Interventions: Combination Product: Laser+clonazepam
- group 2 Laser Sham (Sham Comparator): Group 2 (n=19) were treated with the same laser once a week for a month, but with the tip deactivated
  Interventions: Device: Laser Sham
- group3 laser (Experimental): Group 3 (n=21) were treated with the Helbo® laser once a week for a month.
  Interventions: Device: Laser
- group 4 clonazepam (Experimental): Group 4 (n=18) were treated with Rivotril 0.25mg once a day for a month.
  Interventions: Drug: Clonazepam

INTERVENTIONS:
Combination Product: Laser+clonazepam — treated with the Helbo® Theralite Laser 3D Pocket Probe low power diode laser once a week for a month and Rivotril 0.25mg once every 24 hours for a month
  Arms: Group1 laser + clonazepam
Device: Laser Sham — INACTIVE Helbo® Theralite Laser 3D Pocket Probe low power diode laser once a week for a month
  Arms: group 2 Laser Sham
Device: Laser — Active Helbo® Theralite Laser 3D Pocket Probe low power diode laser once a week for a month
  Arms: group3 laser
Drug: Clonazepam — Rivotril 0.25mg once every 24 hours for a month
  Arms: group 4 clonazepam

SUMMARY:
Burning Mouth Syndrome (BMS) is a chronic pain disorder that presents with inflammation and burning sensation in the oral cavity without visible lesions. Multiple therapies have been investigated without conclusive results.Objective: To analyse the efficacy of treatment with Clonazepam (Rivotril) and Low Power Diode Laser Therapy in patients with Burning Mouth Syndrome and to study the markers of inflammation present in the patients' saliva.

Methods: Randomised, single-blind clinical trial with 89 patients divided into Group 1 Laser + Rivotril (n=20), Group 2 Laser Sham placebo (n=19), Group 3 Laser (n=21) and Group 4 Rivotril (n=18). The intensity of symptomatology was rated by Visual Analogue Scale (VAS). Sialometry was performed before and after treatment and questionnaires such as the Xerostomia Inventory, the Oral Health Impact Profile-14 (OHIP14) and the Mini-Nutritional Assessment (MNA) were completed. Saliva samples were analysed by measuring markers related to inflammatory processes; Interleukins (IL2, IL4, IL 5, IL6, IL 7, IL 8, IL1β, IL 10, IL12, IL13, IL17, IL21, IL23), proteins (MIP-3α, MIP-1α, MIP-1β), Cytokine GM-CSF, Interferon gamma (IFNγ), Interferon Inducible Tα-Cell Chemoattractant (ITAC), Fractalkine and Tumour Necrosis Factor α(TNFα).

DETAILED DESCRIPTION:
Methods: Randomised, single-blind clinical trial with 89 patients divided into Group 1 Laser + Rivotril (n=20), Group 2 Laser Sham placebo (n=19), Group 3 Laser (n=21) and Group 4 Rivotril (n=18). The intensity of symptomatology was rated by Visual Analogue Scale (VAS). Sialometry was performed before and after treatment and questionnaires such as the Xerostomia Inventory, the Oral Health Impact Profile-14 (OHIP14) and the Mini-Nutritional Assessment (MNA) were completed. Saliva samples were analysed by measuring markers related to inflammatory processes; Interleukins (IL2, IL4, IL 5, IL6, IL 7, IL 8, IL1β, IL 10, IL12, IL13, IL17, IL21, IL23), proteins (MIP-3α, MIP-1α, MIP-1β), Cytokine GM-CSF, Interferon gamma (IFNγ), Interferon Inducible Tα-Cell Chemoattractant (ITAC), Fractalkine and Tumour Necrosis Factor α(TNFα).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis Burning Mouth Syndrome (BMS) burning sensation in the oral mucosa or recurrent dysesthetics daily for more than 2 hours a day for more than 3 months, without clinically evident causal lesions

Exclusion Criteria:

* Pregnant or lactating patients
* Oncology patients
* Sjögren's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Pain EVA | Baseline through 1 month
  The intensity of the symptoms was rated using a Visual Analog Scale (VAS) where 0=no pain and 10=maximum possible pain.

SECONDARY OUTCOMES:
salivary biomarkers | Baseline through 1 month
  salivary biomarkers interleukins (IL2, IL4, IL5, IL6, IL7, IL8, IL1β)

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tan HL, Smith JG, Hoffmann J, Renton T. A systematic review of treatment for patients with burning mouth syndrome. Cephalalgia. 2022 Feb;42(2):128-161. doi: 10.1177/03331024211036152. Epub 2021 Aug 18. PMID 34404247
- [Background] Alvarenga-Brant R, Costa FO, Mattos-Pereira G, Esteves-Lima RP, Belem FV, Lai H, Ge L, Gomez RS, Martins CC. Treatments for Burning Mouth Syndrome: A Network Meta-analysis. J Dent Res. 2023 Feb;102(2):135-145. doi: 10.1177/00220345221130025. Epub 2022 Oct 8. PMID 36214096
- [Background] Liu YF, Kim Y, Yoo T, Han P, Inman JC. Burning mouth syndrome: a systematic review of treatments. Oral Dis. 2018 Apr;24(3):325-334. doi: 10.1111/odi.12660. Epub 2017 Mar 30. PMID 28247977